CLINICAL TRIAL: NCT06365073
Title: A Case-control Study on the Clinical Characteristics of 28-day and 90-day Death From Severe Anthrax
Status: Recruiting | Type: Observational
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJIRB20231276
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival group: Patients who survived in 28 days/90 days
- death group: Patients who survived in 28 days/90 days

SUMMARY:
This study is a clinical, multi-center, retrospective, case-control study. Patients clinically diagnosed with severe anthrax who meet the inclusion and exclusion criteria will be included in this study for analysis. Respiratory, circulation, nerve and other vital signs of patients with severe anthrax during hospitalization were recorded, and clinical data such as blood routine, blood biochemistry, coagulation function, myocardial injury, therapeutic drug use, and survival time of patients were recorded, as well as the survival situation of patients 28 days and 90 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. The typical bacilli with capsules were found in smear examination and culture of various secretions, excretions, blood and cerebrospinal fluid.
2. Multiple organ dysfunction (MODS) in brain, heart, liver, kidney, coagulation or more than one organ failure.

Exclusion Criteria:

There are other conditions that affect short-term survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe anthrax
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality rates of severe anthrax | 28 days and 90 days
  mortality rates of severe anthrax

SECONDARY OUTCOMES:
incidence of complications | in hospital
  To evaluate the incidence of respiratory, circulatory, neurological, digestive, coagulation and other complications of severe anthrax
Peripheral blood biomarkers associated with 28-day and 90-day mortality | 28 days and 90 days
  Peripheral blood biomarkers associated with 28-day and 90-day mortality
the improvement in 28-day and 90-day mortality with treatment for severe anthrax | 28 days and 90 days
  the improvement in 28-day and 90-day mortality with treatment for severe anthrax

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China